CLINICAL TRIAL: NCT04355806
Title: A Cohort Study to Evaluate the Impact of Inactivated Trivalent Influenza Vaccine on the Immunogenicity, Safety and Survival of Non-small Cell Lung Cancer Patients Receiving PD-1 / PD-L1 Inhibitors
Brief Title: Impact of Inactivated Trivalent Influenza Vaccine on NSCLC Patients Receiving PD-1 / PD-L1 Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: TIV-NSCLC-PD1
Record Dates: First submitted 2020-04-09; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Non Small Cell Lung Cancer; Influenza Vaccine
Keywords: Non-Small Cell Lung Cancer; Influenza Vaccine; PD-1 Receptor; Programmed Cell Death 1 Ligand 1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Influenza, Human | interventions — Immune Checkpoint Inhibitors; Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen includes the peripheral blood samples collected on day0, 12h, day1, 2, 7, 21, 30, 60 and 6 months after vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaccinated NSCLC group: This group contains 100 NSCLC patients receiving PD-1/PD-L1 inhibitors for more than 6 months, who will be intramuscularly injected one dose of inactivated trivalent influenza vaccine in influenza seasons 2020-21 or 2021-22 (November-May).
  Interventions: Drug: PD-1/PD-L1 inhibitors; Biological: Inactivated trivalent influenza vaccine
- Vaccinated Health group: This group contains 30 healthy participants without immunosuppressive diseases, who will be intramuscularly injected one dose of inactivated trivalent influenza vaccine in influenza seasons 2020-21 or 2021-22 (November-May).
  Interventions: Biological: Inactivated trivalent influenza vaccine
- Unvaccinated NSCLC group: This group contains 30 NSCLC patients receiving PD-1/PD-L1 inhibitors for more than 6 months without intramuscular injection of any inactivated trivalent influenza vaccine in influenza seasons 2020-21 or 2021-22 (November-May).
  Interventions: Drug: PD-1/PD-L1 inhibitors

INTERVENTIONS:
Drug: PD-1/PD-L1 inhibitors — Including nivolumab, pembrolizumab, atezolizumab, and durvalumab, et al.
  Other Names: PD-1/PD-L1 blockades; PD-1 monoclonal antibodies; PD-L1 monoclonal antibodies
  Groups: Unvaccinated NSCLC group; Vaccinated NSCLC group
Biological: Inactivated trivalent influenza vaccine — Including two type A viruses, H1N1 and H3N2, and one type B virus, B/Brisbane.
  Other Names: Flu Vaccines; Influenza Virus Vaccines; Influenza Vaccine, Trivalent; Vaccine, Trivalent Influenza; Flu Shot
  Groups: Vaccinated Health group; Vaccinated NSCLC group

SUMMARY:
This project is to assess the immunogenicity, safety and overall survival impact of intramuscular injection of trivalent influenza vaccine in non-small cell lung cancer (NSCLC) patients with PD-1/PD-L1 inhibitor treatment.

DETAILED DESCRIPTION:
Lung cancer is one of the most prevalent cancers in the world. Among them, non-small cell lung cancer (NSCLC) accounts for about 85%. Immune checkpoint inhibitors such as programmed death 1(PD-1) and PD-L1 are new treatments for NSCLC. About 290,000 to 650,000 people die from respiratory illnesses caused by seasonal flu all over the world. Cancer patients are one of the high-risk groups of influenza. Although the United States, Britain, Australia have issued guidelines recommending that cancer patients be vaccinated against influenza every year, due to concerns about the immune effect and safety of flu vaccination for cancer patients, multiple countries including China have not included cancer patients into priority influenza vaccination populations. Therefore, how to further prove the immunogenicity and safety of influenza vaccine in NSCLC patients is the key to promote influenza vaccines in NSCLC patients.

This study will recruit 130 patients with NSCLC who have been treated with PD-1 / PD-L1 inhibitors for 6 months or more and 30 healthy participants. Among them, 100 NSCLC patients and 30 healthy participants will be intramuscularly inactivated with a trivalent influenza vaccine during the influenza seasons 2020-21 and 2021-22. Vaccinated participants' peripheral blood samples were collected at day0, 12 hours, day1, 2, 7, 21, 30, 60 and 6 months after vaccination. The influenza specific antibody titers, inflammatory chemokines and cytokines, antibody-dependent cellular cytotoxicity (ADCC) activity, T lymphocytes activity and the proportions of different T cells subgroups will be measured to evaluate the participants' immune response to the vaccine. In addition, for the subjects receiving the vaccine, the study will also group by age to compare the differences in immune effects between subjects aged 18-65 and subjects over 65.

At last, this project will compare immune-related adverse events (irAEs) that occurred after receiving PD-1 / PD-L1 inhibitor therapy and survival time between NSCLC patients who receive influenza vaccine and those who do not receive influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. NSCLC patients were diagnosed with clear pathological classification and receive PD-1 / PD-L1 inhibitor treatment during this project.
2. NSCLC patients have the exact start and end time of PD-1 / PD-L1 inhibitor and / or the vaccination time and follow-up information.
3. The healthy participants are not in an immunosuppressive state, such as cancer, HIV, autoimmune diseases, and long-term use of immunosuppressive drugs.
4. The healthy participants have exact vaccination time.
5. All participants have complete clinical and laboratory diagnostic data.
6. All participants are 18-75 years, regardless of gender.
7. All participants have agreed and signed the consent form before enrollment.

Exclusion Criteria:

1. Patients with unclear diagnosis of lung cancer were excluded.
2. Patients with incomplete clinical data or incomplete follow-up records.
3. Patients without signed informed consent.
4. Patient has received blood transfusion within three months.
5. Patients with HIV, Hepatitis B and Hepatitis C infections.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NSCLC patients receiving PD-1/PD-L1 inhibitors during this project
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Titers of anti-nucleoprotein(NP) or anti-hemagglutinin(HA) antibody (IgG and IgM) | Day 0 after vaccination
  The titers of anti-HA IgG and IgM antibodies ,and anti-NP IgG and IgM antibodies are measured by enzyme linked immunosorbent assay (ELISA).
Titers of anti-nucleoprotein(NP) or anti-hemagglutinin(HA) antibody (IgG and IgM) | Day 2 after vaccination
  The titers of anti-HA IgG and IgM antibodies ,and anti-NP IgG and IgM antibodies are measured by enzyme linked immunosorbent assay (ELISA).
Titers of anti-nucleoprotein(NP) or anti-hemagglutinin(HA) antibody (IgG and IgM) | Day 7 after vaccination
  The titers of anti-HA IgG and IgM antibodies ,and anti-NP IgG and IgM antibodies are measured by enzyme linked immunosorbent assay (ELISA).
Titers of anti-nucleoprotein(NP) or anti-hemagglutinin(HA) antibody (IgG and IgM) | Day 21 after vaccination
  The titers of anti-HA IgG and IgM antibodies ,and anti-NP IgG and IgM antibodies are measured by enzyme linked immunosorbent assay (ELISA).
Titers of anti-nucleoprotein(NP) or anti-hemagglutinin(HA) antibody (IgG and IgM) | Day 30 after vaccination
  The titers of anti-HA IgG and IgM antibodies ,and anti-NP IgG and IgM antibodies are measured by enzyme linked immunosorbent assay (ELISA).
Titer of neutralization antibody | Day 0 after vaccination
  Titer of neutralization antibody is measured by neutralization test.
Titer of neutralization antibody | Day 21 after vaccination
  Titer of neutralization antibody is measured by neutralization test.
Titer of neutralization antibody | Day 30 after vaccination
  Titer of neutralization antibody is measured by neutralization test.
Titer of neutralization antibody | Day 60 after vaccination
  Titer of neutralization antibody is measured by neutralization test.
Titer of neutralization antibody | Month 6 after vaccination
  Titer of neutralization antibody is measured by neutralization test.
Multiple chemokine and cytokine levels in peripheral blood | Day 0 after vaccination
  IFN-γ, IL-1β, IL-2,IL-3,IL-4,IL-5,IL-6,IL-8 (CXCL8),IL-9,IL-10,IL-11,IL-12,IL-13,GM-CSF,TNF-α, IP-10 (CXCL10), MCP-1 (CCL2), and TARC (CCL17) in peripheral blood are measured by cytometry bead assay.
Multiple chemokine and cytokine levels in peripheral blood | 12 hours after vaccination
  IFN-γ, IL-1β, IL-2,IL-3,IL-4,IL-5,IL-6,IL-8 (CXCL8),IL-9,IL-10,IL-11,IL-12,IL-13,GM-CSF,TNF-α, IP-10 (CXCL10), MCP-1 (CCL2), and TARC (CCL17) in peripheral blood are measured by cytometry bead assay.
Multiple chemokine and cytokine levels in peripheral blood | Day 1 after vaccination
  IFN-γ, IL-1β, IL-2,IL-3,IL-4,IL-5,IL-6,IL-8 (CXCL8),IL-9,IL-10,IL-11,IL-12,IL-13,GM-CSF,TNF-α, IP-10 (CXCL10), MCP-1 (CCL2), and TARC (CCL17) in peripheral blood are measured by cytometry bead assay.
Multiple chemokine and cytokine levels in peripheral blood | Day 2 after vaccination
  IFN-γ, IL-1β, IL-2,IL-3,IL-4,IL-5,IL-6,IL-8 (CXCL8),IL-9,IL-10,IL-11,IL-12,IL-13,GM-CSF,TNF-α, IP-10 (CXCL10), MCP-1 (CCL2), and TARC (CCL17) in peripheral blood are measured by cytometry bead assay.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | Day 0 after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | 12 hours after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | Day 1 after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | Day 2 after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | Day 7 after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | Day 21 after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | Day 30 after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | Day 60 after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
The numbers and proportions of T lymphocyte subpopulations in peripheral blood | Month 6 after vaccination
  The numbers and proportions of CD4+ T cells, CD8+ T cells, naïve T cells and effector memory T cells in peripheral blood are measured by multiple flow cytometry.
Peripheral T cell activation and proliferation | Day 0 after vaccination
  The CD3, CD4, CD8 and CD69 expressions and cell count of peripheral T cells are measured by multiple flow cytometry upon carboxyfluorescein succinimidyl amino ester (CFSE) labeling and anti-CD3/28 beads activation.
Peripheral T cell activation and proliferation | Day 30 after vaccination
  The CD3, CD4, CD8 and CD69 expressions and cell count of peripheral T cells are measured by multiple flow cytometry upon carboxyfluorescein succinimidyl amino ester (CFSE) labeling and anti-CD3/28 beads activation.
Peripheral T cell activation and proliferation | Day 60 after vaccination
  The CD3, CD4, CD8 and CD69 expressions and cell count of peripheral T cells are measured by multiple flow cytometry upon carboxyfluorescein succinimidyl amino ester (CFSE) labeling and anti-CD3/28 beads activation.
Peripheral T cell activation and proliferation | Month 6 after vaccination
  The CD3, CD4, CD8 and CD69 expressions and cell count of peripheral T cells are measured by multiple flow cytometry upon carboxyfluorescein succinimidyl amino ester (CFSE) labeling and anti-CD3/28 beads activation.
Antibody-dependent cellular cytotoxicity (ADCC) | Day 0 after vaccination
  The ADCC activities of NK-92 cells cultured by the sera from vaccinated participants are measured by lactic acid dehydrogenase (LDH) release of A549 cells infected by H1N1 and H3N2.
Antibody-dependent cellular cytotoxicity (ADCC) | Day 30 after vaccination
  The ADCC activities of NK-92 cells cultured by the sera collected from vaccinated participants are measured by lactic acid dehydrogenase (LDH) release of A549 cells infected by H1N1 and H3N2.
Antibody-dependent cellular cytotoxicity (ADCC) | Day 60 after vaccination
  The ADCC activities of NK-92 cells cultured by the sera collected from vaccinated participants are measured by lactic acid dehydrogenase (LDH) release of A549 cells infected by H1N1 and H3N2.
Antibody-dependent cellular cytotoxicity (ADCC) | Month 6 after vaccination
  The ADCC activities of NK-92 cells cultured by the sera collected from vaccinated participants are measured by lactic acid dehydrogenase (LDH) release of A549 cells infected by H1N1 and H3N2.
Immune-related adverse events (irAEs) | June 2020- June 2023
  The performances and the grades of irAEs according to Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0) and their correlation with vaccination.
Progression-free Survival (PFS) | June 2020- June 2023 (3 year)
  PFS is calculated as the time from from PD-1/PD-L1 inhibitor starting to the disease progression or the death from any cause.
Overall Survival (OS) | June 2020- June 2023 (3 year)
  OS is calculated as the time from PD-1/PD-L1 inhibitor starting to the death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | June 2020- June 2023 (3 year)
  The proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including cases of complete response (CR) and partial response (PR) according to Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1).
Disease Control Rate (DCR) | June 2020- June 2023 (3 year)
  The proportion of patients achieve CR or PR or stable disease (SD) after PD-1/PD-L1 inhibitor treatment according to RECIST 1.1.
Time to Treatment Failure (TFF) | June 2020- June 2023 (3 year)
  The time from the start of PD-1/PD-L1 inhibitor to the withdrawal of the trial. The reasons for withdrawal include the patient's voluntary withdrawal, disease progression, adverse events and even deaths.

CONTACTS AND LOCATIONS:
Overall Officials: Yayi He, PhD, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (2):
- China (2):
  - School of Public Health, Li Ka Shing Faculty of Medicine, University of Hong Kong, Hong Kong, Hong Kong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided